CLINICAL TRIAL: NCT03058692
Title: A Phase II, Double-Blind, Multicenter, Randomized, Placebo-Controlled Trial to Assess the Safety, Reactogenicity and Immunogenicity of Two Doses of Multimeric-001 (M-001) Followed by Seasonal Quadrivalent Influenza Vaccine
Brief Title: Two Doses of Multimeric-001 (M-001) Followed by Influenza Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 14-0112; HHSN272201300015I
Record Dates: First submitted 2017-02-09; First posted 2017-02-23 (Actual); Results first posted 2020-02-05 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2019-11-27

CONDITIONS: Influenza; Influenza Immunisation
Keywords: Immunogenicity; Influenza Vaccine; M-001 vaccine; Reactogenicity; Safety
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- M-001 + IIV4 (Experimental): 0.4 ml injection of M-001 (1 mg dose) intramuscularly on Day 1 and Day 22, followed by 0.5 ml injection of IIV4 (60 mcg HA) intramuscularly on Day 172 (n=60)
  Interventions: Biological: Influenza Multimeric-001 Vaccine; Biological: Quadrivalent Recombinant Seasonal Influenza Vaccine
- Placebo+ IIV4 (Placebo Comparator): 0.4 ml injection of placebo intramuscularly on Day 1 and Day 22, followed by 0.5 ml injection of IIV4 (60 mcg HA) intramuscularly on Day 172 (n=60)
  Interventions: Other: Placebo; Biological: Quadrivalent Recombinant Seasonal Influenza Vaccine

INTERVENTIONS:
Biological: Influenza Multimeric-001 Vaccine — The M-001 vaccine consists of 3 repetitions of 9 conserved linear epitopes that are prepared as a single recombinant protein. The M-001 vaccine is expected to protect against existing as well as future seasonal and pandemic virus strains.
  Arms: M-001 + IIV4
Other: Placebo — Placebo is saline injection
  Arms: Placebo+ IIV4
Biological: Quadrivalent Recombinant Seasonal Influenza Vaccine — Quadrivalent Inactivated Influenza Vaccine (IIV4) for intramuscular injection is indicated for active immunization against influenza disease caused by influenza virus subtypes A and type B present in the vaccine.

SUMMARY:
This is a Phase II randomized, double-blind, placebo-controlled trial in 120 males and non-pregnant females, 18 to 49 years old, inclusive, who are in good health and meet all eligibility criteria. This clinical trial will be conducted at 3 United States sites and is designed to assess the safety, reactogenicity, and immunogenicity of two priming doses of M-001 followed by a seasonal quadrivalent inactivated influenza vaccine (IIV4). The duration of this trial for each subject will be approximately 7 months. The entire study duration will be approximately 24 months. The primary objectives are: 1) To assess the safety as measured by vaccine related adverse events, reactogenicity, and laboratory adverse events of two doses of M-001 vaccine, each dose administered approximately 21 days apart; and 2) To assess the T cell responses to M-001 component peptides following two doses of M-001.

DETAILED DESCRIPTION:
This is a Phase II randomized, double-blind, placebo-controlled trial in 120 males and non-pregnant females, 18 to 49 years old, inclusive, who are in good health and meet all eligibility criteria. This clinical trial will be conducted at 3 United States sites and is designed to assess the safety, reactogenicity, and immunogenicity of two priming doses of M-001 followed by a seasonal quadrivalent inactivated influenza vaccine (IIV4). The duration of this trial for each subject will be approximately 7 months. The entire study duration will be approximately 24 months. The primary objectives are: 1) To assess the safety as measured by vaccine related adverse events, reactogenicity, and laboratory adverse events of two doses of M-001 vaccine, each dose administered approximately 21 days apart; and 2) To assess the T cell responses to M-001 component peptides following two doses of M-001. The secondary objectives are: 1) To assess all serious adverse events (SAEs) following receipt of each dose of M-001 vaccine or placebo, each dose separated by approximately 21 days, through the end of the study; 2) To assess all unsolicited non-serious AEs following receipt of each dose of M-001 or placebo, each dose separated by approximately 21 days, through 21 days after each dose of M-001 or placebo; and 3) To assess the serum HAI and Neut antibody responses to the 2018-2019 IIV4 vaccine viruses.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent prior to initiation of any study procedures.
2. Are able to understand and comply with planned study procedures and be available for all study visits.
3. Are males or non-pregnant females, 18 to 49 years old, inclusive.
4. Are in good health*.

   *As determined by medical history and targeted physical examination to evaluate acute or currently ongoing chronic medical diagnoses or conditions, defined as those that have been present for at least 90 days, which would affect the assessment of the safety of subjects or the immunogenicity of study vaccinations. Chronic medical diagnoses or conditions should be stable for the last 60 days prior to investigational vaccine study product administration. This includes no change in chronic prescription medication, dose, or frequency as a result of deterioration of the chronic medical diagnosis or condition in the 60 days prior to enrollment and investigational vaccine study product administration. Any prescription change that is due to change of health care provider, insurance company, etc., or that is done for financial reasons, as long as in the same class of medication, will not be considered a deviation of this inclusion criterion. Any change in prescription medication due to improvement of a disease outcome, as determined by the site principal investigator or appropriate sub-investigator, will not be considered a deviation of this inclusion criterion. Subjects may be on chronic or as needed (prn) medications if, in the opinion of the site principal investigator or appropriate sub-investigator, they pose no additional risk to subject safety or assessment of reactogenicity and immunogenicity and do not indicate a worsening of medical diagnosis or condition. Similarly, medication changes subsequent to enrollment and investigational study product vaccination are acceptable provided there was no deterioration in the subject's chronic medical condition that necessitated a medication change. All chronic medical condtions should pose no additional risk to the subject or interference with the evaluation of responses to study vaccination. Note: Topical, nasal, and inhaled medications (with the exception of inhaled corticosteroids as outlined in the Subject Exclusion Criteria), herbals, vitamins, and supplements are permitted.
5. Oral temperature is less than 100.0 degrees F.
6. Pulse** is 50 to 100 bpm, inclusive.

   **Acceptable pulse range prior to IIV4 dose is 45 to 115 bpm, inclusive and no symptoms.
7. Systolic blood pressure*** is 85 to 150 mmHg, inclusive. ***Acceptable systolic blood pressure range prior to IIV4 dose is 80 to 155 mm Hg, inclusive and no symptoms.
8. Diastolic blood pressure**** is 55 to 95 mmHg, inclusive.

   ****Acceptable diastolic blood pressure range prior to IIV4 dose is 50 to 100 mm Hg, inclusive and no symptoms.
9. Women of childbearing potential* must use an acceptable method of contraception** from 30 days prior to vaccination until 60 days after the second of dose of M-001 or placebo.
10. Women of childbearing potential***** must use an acceptable method of contraception****** from 30 days prior to receipt of IIV vaccination, and must plan to use until 28 days after the IIV.

    *****Not sterilized via tubal ligation, bilateral oophorectomy, hysterectomy, or successful Essure(R) placement (permanent, non-surgical, non-hormonal sterilization with history of documented radiological confirmation test achieved or with use of another approved birth control method if confirmation test not confirmed) and still menstruating or < 1 year of the last menses if menopausal).

    ******Includes, but is not limited to, non-male sexual relationships, abstinence from sexual intercourse with a male partner, monogamous relationship with a vasectomized partner, male condoms with the use of applied spermicide, intrauterine devices, NuvaRing(R), and licensed hormonal methods such as implants, injectables, contraceptive patches or oral contraceptives ("the pill"). Method of contraception will be captured on the appropriate data collection form.
11. Female subjects of childbearing potential must have a negative urine or serum pregnancy test within 24 hours prior to study vaccination.

Exclusion Criteria:

1. Have an acute illness*, as determined by the site PI or appropriate sub-investigator, within 72 hours prior to study vaccination.

   * An acute illness which is nearly resolved with only minor residual symptoms remaining is allowable if, in the opinion of the site PI or appropriate sub-investigator, the residual symptoms will not interfere with the ability to assess safety parameters as required by the protocol.
2. Have any medical disease or condition that, in the opinion of the site PI or appropriate sub-investigator, is a contraindication to study participation**.

   **Including acute or chronic medical disease or condition, defined as persisting for at least 90 days, that would place the subject at an unacceptable risk of injury, render the subject unable to meet the requirements of the protocol, or may interfere with the evaluation of responses or the subject's successful completion of this study.
3. Have immunosuppression as a result of an underlying illness or treatment, or use of anticancer chemotherapy or radiation therapy (cytotoxic) within 3 years prior to study vaccination.
4. Have known active neoplastic disease or a history of any hematologic malignancy. Non-melanoma skin cancers that are not active are permitted.
5. Have known HIV, hepatitis B, or hepatitis C infection.
6. Have known hypersensitivity or allergy to eggs, egg or chicken protein, or other components of the study vaccine.
7. Have a history of severe reactions following previous immunization with licensed or unlicensed influenza vaccines.
8. Have a history of Guillain-Barré Syndrome.
9. Have a history of alcohol or drug abuse within 5 years prior to study vaccination.
10. Have any diagnosis, current or past, of schizophrenia, bipolar disease, or other psychiatric diagnosis that may interfere with subject compliance or safety evaluations.
11. Have been hospitalized for psychiatric illness, history of suicide attempt, or confinement for danger to self or others within 10 years prior to study vaccination.
12. Have taken oral or parenteral (including intraarticular) corticosteroids of any dose within 30 days prior to study vaccination.
13. Have taken high-dose*** dose inhaled corticosteroids within 30 days prior to study vaccination****.

    ***High-dose defined as per age as using inhaled high dose per reference chart https://www.nhlbi.nih.gov/health-pro/guidelines/current/asthma-guidelines/quick-reference-html#estimated-comparative-daily-doses.

    ****Topical and nasal steroids are permissible.
14. Received any licensed live vaccine or plan to receive a licensed live vaccine within 30 days prior or 21 days after each M-001 study vaccination.
15. Received a licensed inactivated vaccine within 14 days prior to or 21 days after each M-001 study vaccination.
16. Plans to or received the current 2018-2019 influenza vaccine (inactivated or live prior to ordering the study (the 2018-2019 influenza vaccine will be given during the trial.))
17. Received immunoglobulin or other blood products (with exception of Rho D immunoglobulin) within 90 days prior to study vaccination.
18. Received an experimental agent***** within 30 days prior to the first study vaccination, or expects to receive an experimental agent****** during the 7-month trial-reporting period.

    *****Including vaccine, drug, biologic, device, blood product, or medication.

    ******Other than from participation in this study.
19. Are participating or plan to participate in another clinical trial with an interventional agent******* that will be received during the 7-month trial-reporting period.

    *******Including agent (licensed or unlicensed vaccine, drug, biologic, device, blood product, or medication) during the 9-month study period.
20. Plan to travel outside the U.S. (continental U.S., Hawaii and Alaska) in the time between the first study vaccination and 21 days after the last study vaccination********.

    ********Study vaccination refers to investigational study product vaccination.
21. Female subjects who are breastfeeding or plan to breastfeed at any given time from the first study vaccination until 30 days after the last study vaccination.
22. Blood donation or planned blood donation within 30 days prior to the study vaccination through 30 days after the last blood drawn for this study.
23. Have signs or symptoms that could confound or confuse assessment of study vaccine reactogenicity*********.

    *********The study vaccination should be postponed/deferred until signs or symptoms have resolved and if within the acceptable protocol-specified window for that visit.
24. Have a history of convulsions or encephalomyelitis within 90 days prior to study vaccination.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2019-01-14 (Actual); Study Completion 2019-01-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Iowa - Vaccine Research and Education Unit, Iowa City, Iowa
  - Cincinnati Children's Hospital Medical Center - Infectious Diseases, Cincinnati, Ohio
  - Baylor College of Medicine - Molecular Virology and Microbiology, Houston, Texas

REFERENCES:
- [Derived] Atmar RL, Bernstein DI, Winokur P, Frey SE, Angelo LS, Bryant C, Ben-Yedidia T, Roberts PC, El Sahly HM, Keitel WA. Safety and immunogenicity of Multimeric-001 (M-001) followed by seasonal quadrivalent inactivated influenza vaccine in young adults - A randomized clinical trial. Vaccine. 2023 Apr 17;41(16):2716-2722. doi: 10.1016/j.vaccine.2023.03.023. Epub 2023 Mar 21. PMID 36941155

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were healthy adult males and non-pregnant females recruited from existing volunteer populations and from the communities at large around the clinical sites. Participants were enrolled between 09APR2018 and 28JUN2018.
Groups:
- M-001 + IIV4: 0.4 ml injection of M-001 (1 mg dose) intramuscularly on Day 1 and Day 22, followed by 0.5 ml injection of IIV4 (60 mcg HA) intramuscularly on Day 172
  Influenza Multimeric-001 Vaccine: The M-001 vaccine consists of 3 repetitions of 9 conserved linear epitopes that are prepared as a single recombinant protein. The M-001 vaccine is expected to protect against existing as well as future seasonal and pandemic virus strains.
  Quadrivalent Recombinant Seasonal Influenza Vaccine: Quadrivalent Inactivated Influenza Vaccine (IIV4) for intramuscular injection is indicated for active immunization against influenza disease caused by influenza virus subtypes A and type B present in the vaccine.
- Placebo + IIV4: 0.4 ml injection of placebo intramuscularly on Day 1 and Day 22, followed by 0.5 ml injection of IIV4 (60 mcg HA) intramuscularly on Day 172
  Placebo: Placebo is saline injection
  Quadrivalent Recombinant Seasonal Influenza Vaccine: Quadrivalent Inactivated Influenza Vaccine (IIV4) for intramuscular injection is indicated for active immunization against influenza disease caused by influenza virus subtypes A and type B present in the vaccine.
Period: Overall Study
Arm/Group | M-001 + IIV4 | Placebo + IIV4
Started | 61 | 59
Completed | 58 | 57
Not Completed | 3 | 2
Not completed — Lost to Follow-up | 2 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: The baseline analysis population includes all subjects.
Groups:
- M-001 + IIV4: 0.4 ml (1 mg) M-001 IM on Day 1 and Day 22, followed by 0.5 ml IIV4 IM on Day 172
- Placebo + IIV4: 0.4 ml Placebo IM on Day 1 and Day 22, followed by 0.5 ml IIV4 IM on Day 172
- Total: Total of all reporting groups
Arm/Group | M-001 + IIV4 | Placebo + IIV4 | Total
Number analyzed (Participants) | 61 | 59 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 61 | 59 | 120
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.6 (7.9) | 33.5 (7.8) | 33.0 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 33 | 75
  Male | 19 | 26 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 6 | 11
  Not Hispanic or Latino | 56 | 53 | 109
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 8 | 5 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 49 | 50 | 99
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 61 | 59 | 120

OUTCOME MEASURES:

1. Primary Outcome: Mean Percentage of Perforin+ CD4+ and CD8+ T Cells After Stimulation With M-001 Component Peptides
Description: The percentages of CD4 and CD8 T cells expressing markers were determined using fluorescence-based flow cytometric assays from cryopreserved PBMCs collected and isolated from participants at Day 1 prior to initial vaccination and again at 14 days after the second vaccination. The percentages were calculated as the number of cells positive for these proteins divided by the total number of CD4+ or CD8+ T cells counted in each sample.
Time Frame: Day 1 through Day 36
Population: The modified intent-to-treat (mITT) population includes all subjects who received at least one dose of study vaccine and contributed at least one post-study vaccination venous blood sample for immunogenicity testing for which valid results were reported.
Measure: Mean (95% Confidence Interval); unit: percentage of cells
Arm/Group | M-001 + IIV4 | Placebo + IIV4
Number analyzed (Participants) | 58 | 59
percentage of cells
  Perforin+ CD4+ at Day 1 | 1.180 [0.724 to 1.700] | 0.781 [0.464 to 1.140]
  Perforin+ CD4+ Day 36 | 1.090 [0.649 to 1.610] | 0.779 [0.470 to 1.140]
  Perforin+ CD8+ Day 1 | 16.1 [12.9 to 19.4] | 12.4 [10.4 to 14.5]
  Perforin+ CD8+ Day 36 | 16.3 [13.1 to 19.7] | 13.8 [11.4 to 16.3]
Statistical Analysis 1: Comparison: M-001 + IIV4 vs Placebo + IIV4; This reports the analysis for response in CD4+ T cells at Day 36. The null hypothesis for the non-parametric test assumed both groups are from the same population, i.e., are homogeneous and have the same distribution. The study was not designed/powered to detect differences between groups in the frequencies of marker combinations, considering the issue of multiplicity; Test type: Other; p = 0.53, Wilcoxon (Mann-Whitney) — As this trial was not confirmatory, as common for early phase trials, p-values were not adjusted for multiple comparisons, rather included to aid interpretation of the estimates. A priori threshold for statistical significance was not defined
Statistical Analysis 2: Comparison: M-001 + IIV4 vs Placebo + IIV4; This reports the analysis for response in CD8+ T cells at Day 36. The null hypothesis for the non-parametric test assumed both groups are from the same population, i.e., are homogeneous and have the same distribution. The study was not designed/powered to detect differences between groups in the frequencies of marker combinations, considering the issue of multiplicity; Test type: Other; p = 0.56, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

2. Primary Outcome: Mean Percentage of Cluster of Differentiation 107a Positive (CD107a+) CD4+ and CD8+ T Cells After Stimulation With M-001 Component Peptides
Description: as for outcome 1
Time Frame: Day 1 through Day 36
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of cells
Arm/Group | M-001 + IIV4 | Placebo + IIV4
Number analyzed (Participants) | 58 | 59
percentage of cells
  CD107a+ CD4+ at Day 1 | 0.255 [0.195 to 0.323] | 0.264 [0.198 to 0.342]
  CD107a+ CD4+ Day 36 | 0.242 [0.191 to 0.301] | 0.257 [0.205 to 0.317]
  CD107a+ CD8+ Day 1 | 0.348 [0.277 to 0.425] | 0.367 [0.277 to 0.479]
  CD107a+ CD8+ Day 36 | 0.352 [0.283 to 0.428] | 0.384 [0.305 to 0.473]
Statistical Analysis 1: Comparison: M-001 + IIV4 vs Placebo + IIV4; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.74, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: M-001 + IIV4 vs Placebo + IIV4; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.73, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

3. Primary Outcome: Mean Percentage of Interleukin-2 Positive (IL-2+) CD4+ and CD8+ T Cells After Stimulation With M-001 Component Peptides
Description: as for outcome 1
Time Frame: Day 1 through Day 36
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of cells
Arm/Group | M-001 + IIV4 | Placebo + IIV4
Number analyzed (Participants) | 58 | 59
percentage of cells
  IL-2+ CD4+ at Day 1 | 0.0682 [0.0481 to 0.0910] | 0.0634 [0.0503 to 0.0776]
  IL-2+ CD4+ Day 36 | 0.0749 [0.0584 to 0.0930] | 0.0692 [0.0537 to 0.0866]
  IL-2+ CD8+ Day 1 | 0.1260 [0.0789 to 0.1910] | 0.0939 [0.0716 to 0.1180]
  IL-2+ CD8+ Day 36 | 0.1010 [0.0763 to 0.1300] | 0.1170 [0.0883 to 0.1480]
Statistical Analysis 1: Comparison: M-001 + IIV4 vs Placebo + IIV4; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.66, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: M-001 + IIV4 vs Placebo + IIV4; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.48, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

4. Primary Outcome: Mean Percentage of Tumor Necrosis Factor Positive (TNF+) CD4+ and CD8+ T Cells After Stimulation With M-001 Component Peptides
Description: as for outcome 1
Time Frame: Day 1 through Day 36
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of cells
Arm/Group | M-001 + IIV4 | Placebo + IIV4
Number analyzed (Participants) | 58 | 59
percentage of cells
  TNF+ CD4+ at Day 1 | 0.437 [0.321 to 0.567] | 0.530 [0.366 to 0.733]
  TNF+ CD4+ Day 36 | 0.450 [0.334 to 0.594] | 0.395 [0.296 to 0.509]
  TNF+ CD8+ Day 1 | 0.0750 [0.0492 to 0.1090] | 0.0716 [0.0495 to 0.1000]
  TNF+ CD8+ Day 36 | 0.0676 [0.0431 to 0.1060] | 0.0596 [0.0437 to 0.0783]
Statistical Analysis 1: Comparison: M-001 + IIV4 vs Placebo + IIV4; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.32, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: M-001 + IIV4 vs Placebo + IIV4; [analysis description as in outcome 1, analysis 1]; Test type: Other; p > 0.99, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

5. Primary Outcome: Mean Percentage of Interferon Gamma Positive (IFNg+) CD4+ and CD8+ T Cells After Stimulation With M-001 Component Peptides
Description: as for outcome 1
Time Frame: Day 1 through Day 36
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of cells
Arm/Group | M-001 + IIV4 | Placebo + IIV4
Number analyzed (Participants) | 58 | 59
percentage of cells
  INFg+ CD4+ at Day 1 | 0.0418 [0.0329 to 0.0532] | 0.0333 [0.0274 to 0.0406]
  INFg+ CD4+ Day 36 | 0.0512 [0.0419 to 0.0621] | 0.0436 [0.0298 to 0.0654]
  INFg+ CD8+ Day 1 | 0.0558 [0.0345 to 0.0843] | 0.0400 [0.0289 to 0.0546]
  INFg+ CD8+ Day 36 | 0.0529 [0.0377 to 0.0709] | 0.0476 [0.0341 to 0.0643]
Statistical Analysis 1: Comparison: M-001 + IIV4 vs Placebo + IIV4; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.0078, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: M-001 + IIV4 vs Placebo + IIV4; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.94, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

6. Primary Outcome: Mean Percentage of Perforin+CD107a+IL-2+TNF+IFNg+ CD4+ and CD8+ T Cells After Stimulation With M-001 Component Peptides
Description: as for outcome 1
Time Frame: Day 1 through Day 36
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of cells
Arm/Group | M-001 + IIV4 | Placebo + IIV4
Number analyzed (Participants) | 58 | 59
percentage of cells
  Perforin+CD107a+IL-2+TNF+IFNg+ CD4+ at Day 1 | 0 [NA to NA] — Not calculable, no cells positive for markers | 0.000067 [0 to 0.000174]
  Perforin+CD107a+IL-2+TNF+IFNg+ CD4+ Day 36 | 0 [NA to NA] — Not calculable, no cells positive for markers | 0 [NA to NA] — Not calculable, no cells positive for markers
  Perforin+CD107a+IL-2+TNF+IFNg+ CD8+ Day 1 | 0 [NA to NA] — Not calculable, no cells positive for markers | 0 [NA to NA] — Not calculable, no cells positive for markers
  Perforin+CD107a+IL-2+TNF+IFNg+ CD8+ Day 36 | 0.0000698 [0 to 0.000209] | 0 [NA to NA] — Not calculable, no cells positive for markers
Statistical Analysis 1: Comparison: M-001 + IIV4 vs Placebo + IIV4; [analysis description as in outcome 1, analysis 1]; Test type: Other; No non-zero results were reported for either group so statistical testing was not performed
Statistical Analysis 2: Comparison: M-001 + IIV4 vs Placebo + IIV4; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.5, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

7. Primary Outcome: Mean Percentage of Perforin+CD107a+IL-2+TNF+IFNg- CD4+ and CD8+ T Cells After Stimulation With M-001 Component Peptides
Description: as for outcome 1
Time Frame: Day 1 through Day 36
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of cells
Arm/Group | M-001 + IIV4 | Placebo + IIV4
Number analyzed (Participants) | 58 | 59
percentage of cells
  Perforin+CD107a+IL-2+TNF+IFNg- CD4+ Day 1 | 0 [NA to NA] — Not calculable, no cells positive for markers | 0 [NA to NA] — Not calculable, no cells positive for markers
  Perforin+CD107a+IL-2+TNF+IFNg- CD4+ Day 36 | 0 [NA to NA] — Not calculable, no cells positive for markers | 0 [NA to NA] — Not calculable, no cells positive for markers
  Perforin+CD107a+IL-2+TNF+IFNg- CD8+ Day 1 | 0 [NA to NA] — Not calculable, no cells positive for markers | 0 [NA to NA] — Not calculable, no cells positive for markers
  Perforin+CD107a+IL-2+TNF+IFNg- CD8+ Day 36 | 0 [NA to NA] — Not calculable, no cells positive for markers | 0 [NA to NA] — Not calculable, no cells positive for markers
Statistical Analysis 1: Comparison: M-001 + IIV4 vs Placebo + IIV4; [analysis description as in outcome 1, analysis 1]; Test type: Other; No non-zero results were reported for either group so statistical testing was not performed
Statistical Analysis 2: Comparison: M-001 + IIV4 vs Placebo + IIV4; [analysis description as in outcome 1, analysis 2]; Test type: Other; No non-zero results were reported for either group so statistical testing was not performed

8. Primary Outcome: Mean Percentage of Perforin+CD107a+IL-2+TNF- IFNg+ CD4+ and CD8+ T Cells After Stimulation With M-001 Component Peptides
Description: as for outcome 1
Time Frame: Day 1 through Day 36
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of cells
Arm/Group | M-001 + IIV4 | Placebo + IIV4
Number analyzed (Participants) | 58 | 59
percentage of cells
  Perforin+CD107a+IL-2+TNF- IFNg+ CD4+ Day 1 | 0 [NA to NA] — Not calculable, no cells positive for markers | 0 [NA to NA] — Not calculable, no cells positive for markers
  Perforin+CD107a+IL-2+TNF- IFNg+ CD4+ Day 36 | 0 [NA to NA] — Not calculable, no cells positive for markers | 0 [NA to NA] — Not calculable, no cells positive for markers
  Perforin+CD107a+IL-2+TNF- IFNg+ CD8+ Day 1 | 0 [NA to NA] — Not calculable, no cells positive for markers | 0 [NA to NA] — Not calculable, no cells positive for markers
  Perforin+CD107a+IL-2+TNF- IFNg+ CD8+ Day 36 | 0 [NA to NA] — Not calculable, no cells positive for markers | 0 [NA to NA] — Not calculable, no cells positive for markers
Statistical Analysis 1: Comparison: M-001 + IIV4 vs Placebo + IIV4; [analysis description as in outcome 1, analysis 1]; Test type: Other; No non-zero results were reported for either group so statistical testing was not performed

9. Primary Outcome: Mean Percentage of Perforin+CD107a+IL-2+TNF- IFNg- CD4+ and CD8+ T Cells After Stimulation With M-001 Component Peptides
Description: as for outcome 1
Time Frame: Day 1 through Day 36
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of cells
Arm/Group | M-001 + IIV4 | Placebo + IIV4
Number analyzed (Participants) | 58 | 59
percentage of cells
  Perforin+CD107a+IL-2+TNF- IFNg- CD4+ Day 1 | 0 [NA to NA] — Not calculable, no cells positive for markers | 0 [NA to NA] — Not calculable, no cells positive for markers
  Perforin+CD107a+IL-2+TNF- IFNg- CD4+ Day 36 | 0 [NA to NA] — Not calculable, no cells positive for markers | 0 [NA to NA] — Not calculable, no cells positive for markers
  Perforin+CD107a+IL-2+TNF- IFNg- CD8+ Day 1 | 0.00033 [0 to 0.00078] | 0.0000461 [0 to 0.000138]
  Perforin+CD107a+IL-2+TNF- IFNg- CD8+ Day 36 | 0 [NA to NA] — Not calculable, no cells positive for markers | 0.0001540 [0 to 0.000387]
Statistical Analysis 1: Comparison: M-001 + IIV4 vs Placebo + IIV4; [analysis description as in outcome 1, analysis 1]; Test type: Other; No non-zero results were reported for either group so statistical testing was not performed
Statistical Analysis 2: Comparison: M-001 + IIV4 vs Placebo + IIV4; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.5, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

10. Primary Outcome: Mean Percentage of Perforin+CD107a+IL-2-TNF+IFNg+ CD4+ and CD8+ T Cells After Stimulation With M-001 Component Peptides
Description: as for outcome 1
Time Frame: Day 1 through Day 36
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of cells
Arm/Group | M-001 + IIV4 | Placebo + IIV4
Number analyzed (Participants) | 58 | 59
percentage of cells
  Perforin+CD107a+IL-2-TNF+IFNg+ CD4+ at Day 1 | 0.0000741 [0 to 0.000191] | 0.000107 [0 to 0.000245]
  Perforin+CD107a+IL-2-TNF+IFNg+ CD4+ Day 36 | 0.0001600 [0 to 0.000370] | 0.000344 [0 to 0.000907]
  Perforin+CD107a+IL-2-TNF+IFNg+ CD8+ Day 1 | 0.00271 [0.000636 to 0.00586] | 0.000269 [0 to 0.00062]
  Perforin+CD107a+IL-2-TNF+IFNg+ CD8+ Day 36 | 0.00187 [0.000358 to 0.00384] | 0.00122 [0.000475 to 0.00209]
Statistical Analysis 1: Comparison: M-001 + IIV4 vs Placebo + IIV4; [analysis description as in outcome 1, analysis 1]; Test type: Other; p > 0.99, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: M-001 + IIV4 vs Placebo + IIV4; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.74, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

11. Primary Outcome: Mean Percentage of Perforin+CD107a+IL-2- TNF+IFNg- CD4+ and CD8+ T Cells After Stimulation With M-001 Component Peptides
Description: as for outcome 1
Time Frame: Day 1 through Day 36
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of cells
Arm/Group | M-001 + IIV4 | Placebo + IIV4
Number analyzed (Participants) | 58 | 59
percentage of cells
  Perforin+CD107a+IL-2-TNF+IFNg- CD4+ at Day 1 | 0.000036 [0 to 0.000108] | 0 [NA to NA] — Not calculable, no cells positive for markers
  Perforin+CD107a+IL-2-TNF+IFNg- CD4+ Day 36 | 0 [NA to NA] — Not calculable, no cells positive for markers | 0.000161 [0 to 0.000445]
  Perforin+CD107a+IL-2-TNF+IFNg- CD8+ Day 1 | 0.00288 [0.000972 to 0.00536] | 0.00172 [0.000753 to 0.00294]
  Perforin+CD107a+IL-2-TNF+IFNg- CD8+ Day 36 | 0.00326 [0.001060 to 0.00606] | 0.00134 [0.000606 to 0.00223]
Statistical Analysis 1: Comparison: M-001 + IIV4 vs Placebo + IIV4; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.50, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: M-001 + IIV4 vs Placebo + IIV4; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.90, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

12. Primary Outcome: Mean Percentage of Perforin+CD107a+IL-2-TNF- IFNg+ CD4+ and CD8+ T Cells After Stimulation With M-001 Component Peptides
Description: as for outcome 1
Time Frame: Day 1 through Day 36
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of cells
Arm/Group | M-001 + IIV4 | Placebo + IIV4
Number analyzed (Participants) | 58 | 59
percentage of cells
  Perforin+CD107a+IL-2-TNF- IFNg+ CD4+ at Day 1 | 0 [NA to NA] — Not calculable, no cells positive for markers | 0 [NA to NA] — Not calculable, no cells positive for markers
  Perforin+CD107a+IL-2-TNF- IFNg+ CD4+ Day 36 | 0.0000566 [0 to 0.00017] | 0.000118 [0 to 0.000318]
  Perforin+CD107a+IL-2-TNF- IFNg+ CD8+ Day 1 | 0.000444 [0.0000800 to 0.000959] | 0.000409 [0 to 0.000963]
  Perforin+CD107a+IL-2-TNF- IFNg+ CD8+ Day 36 | 0.000323 [0.0000639 to 0.000672] | 0.000197 [0 to 0.000518]
Statistical Analysis 1: Comparison: M-001 + IIV4 vs Placebo + IIV4; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.87, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: M-001 + IIV4 vs Placebo + IIV4; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.57, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

13. Primary Outcome: Mean Percentage of Perforin+CD107a+IL-2-TNF- IFNg- CD4+ and CD8+ T Cells After Stimulation With M-001 Component Peptides
Description: as for outcome 1
Time Frame: Day 1 through Day 36
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of cells
Arm/Group | M-001 + IIV4 | Placebo + IIV4
Number analyzed (Participants) | 58 | 59
percentage of cells
  Perforin+CD107a+IL-2-TNF- IFNg- CD4+ at Day 1 | 0.00104 [0.000455 to 0.00175] | 0.000728 [0.000330 to 0.00122]
  Perforin+CD107a+IL-2-TNF- IFNg- CD4+ Day 36 | 0.00123 [0.000602 to 0.00199] | 0.000928 [0.000505 to 0.00141]
  Perforin+CD107a+IL-2-TNF- IFNg- CD8+ Day 1 | 0.0317 [0.0249 to 0.0390] | 0.0237 [0.0148 to 0.0363]
  Perforin+CD107a+IL-2-TNF- IFNg- CD8+ Day 36 | 0.0368 [0.0273 to 0.0472] | 0.0263 [0.0171 to 0.0402]
Statistical Analysis 1: Comparison: M-001 + IIV4 vs Placebo + IIV4; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.82, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: M-001 + IIV4 vs Placebo + IIV4; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.076, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

14. Primary Outcome: Mean Percentage of Perforin+CD107a- IL-2+TNF+IFNg+ CD4+ and CD8+ T Cells After Stimulation With M-001 Component Peptides
Description: as for outcome 1
Time Frame: Day 1 through Day 36
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of cells
Arm/Group | M-001 + IIV4 | Placebo + IIV4
Number analyzed (Participants) | 58 | 59
percentage of cells
  Perforin+CD107a- IL-2+TNF+IFNg+ CD4+ at Day 1 | 0.0000621 [0 to 0.000186] | 0.0000457 [0 to 0.000137]
  Perforin+CD107a- IL-2+TNF+IFNg+ CD4+ Day 36 | 0.0000888 [0 to 0.000229] | 0.0001010 [0 to 0.000276]
  Perforin+CD107a- IL-2+TNF+IFNg+ CD8+ Day 1 | 0.000123 [0 to 0.000369] | 0 [NA to NA] — Not calculable, no cells positive for markers
  Perforin+CD107a- IL-2+TNF+IFNg+ CD8+ Day 36 | 0.000184 [0 to 0.000482] | 0.000128 [0 to 0.000333]
Statistical Analysis 1: Comparison: M-001 + IIV4 vs Placebo + IIV4; [analysis description as in outcome 1, analysis 1]; Test type: Other; p > 0.99, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: M-001 + IIV4 vs Placebo + IIV4; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.75, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

15. Primary Outcome: Mean Percentage of Perforin+CD107a- IL-2+TNF+IFNg- CD4+ and CD8+ T Cells After Stimulation With M-001 Component Peptides
Description: as for outcome 1
Time Frame: Day 1 through Day 36
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of cells
Arm/Group | M-001 + IIV4 | Placebo + IIV4
Number analyzed (Participants) | 58 | 59
percentage of cells
  Perforin+CD107a- IL-2+TNF+IFNg- CD4+ at Day 1 | 0.0000375 [0 to 0.0001130] | 0 [NA to NA] — Not calculable, no cells positive for markers
  Perforin+CD107a- IL-2+TNF+IFNg- CD4+ Day 36 | 0.0000327 [0 to 0.0000982] | 0 [NA to NA] — Not calculable, no cells positive for markers
  Perforin+CD107a- IL-2+TNF+IFNg- CD8+ Day 1 | 0.0005150 [0 to 0.001160] | 0.000322 [0 to 0.000966]
  Perforin+CD107a- IL-2+TNF+IFNg- CD8+ Day 36 | 0.0000524 [0 to 0.000157] | 0 [NA to NA] — Not calculable, no cells positive for markers
Statistical Analysis 1: Comparison: M-001 + IIV4 vs Placebo + IIV4; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.50, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: M-001 + IIV4 vs Placebo + IIV4; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.50, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

16. Primary Outcome: Mean Percentage of Perforin+CD107a- IL-2+TNF- IFNg+ CD4+ and CD8+ T Cells After Stimulation With M-001 Component Peptides
Description: as for outcome 1
Time Frame: Day 1 through Day 36
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of cells
Arm/Group | M-001 + IIV4 | Placebo + IIV4
Number analyzed (Participants) | 58 | 59
percentage of cells
  Perforin+CD107a- IL-2+TNF- IFNg+ CD4+ at Day 1 | 0 [NA to NA] — Not calculable, no cells positive for markers | 0.000101 [0 to 0.000303]
  Perforin+CD107a- IL-2+TNF- IFNg+ CD4+ Day 36 | 0 [NA to NA] — Not calculable, no cells positive for markers | 0.000061 [0 to 0.000183]
  Perforin+CD107a- IL-2+TNF- IFNg+ CD8+ Day 1 | 0 [NA to NA] — Not calculable, no cells positive for markers | 0.0003780 [0 to 0.00113]
  Perforin+CD107a- IL-2+TNF- IFNg+ CD8+ Day 36 | 0 [NA to NA] — Not calculable, no cells positive for markers | 0.0000966 [0 to 0.00029]
Statistical Analysis 1: Comparison: M-001 + IIV4 vs Placebo + IIV4; [analysis description as in outcome 1, analysis 1]; Test type: Other; p > .99, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: M-001 + IIV4 vs Placebo + IIV4; [analysis description as in outcome 1, analysis 2]; Test type: Other; p > .99, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

17. Primary Outcome: Mean Percentage of Perforin+CD107a- IL-2+TNF- IFNg- CD4+ and CD8+ T Cells After Stimulation With M-001 Component Peptides
Description: as for outcome 1
Time Frame: Day 1 through Day 36
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of cells
Arm/Group | M-001 + IIV4 | Placebo + IIV4
Number analyzed (Participants) | 58 | 59
percentage of cells
  Perforin+CD107a- IL-2+TNF- IFNg- CD4+ at Day 1 | 0.00399 [0.00211 to 0.00635] | 0.00307 [0.00134 to 0.00550]
  Perforin+CD107a- IL-2+TNF- IFNg- CD4+ Day 36 | 0.00458 [0.00216 to 0.00748] | 0.00354 [0.00201 to 0.00530]
  Perforin+CD107a- IL-2+TNF- IFNg- CD8+ Day 1 | 0.0742 [0.0385 to 0.1300] | 0.0434 [0.0315 to 0.0568]
  Perforin+CD107a- IL-2+TNF- IFNg- CD8+ Day 36 | 0.0546 [0.0398 to 0.0731] | 0.0612 [0.0417 to 0.0841]
Statistical Analysis 1: Comparison: M-001 + IIV4 vs Placebo + IIV4; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.81, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: M-001 + IIV4 vs Placebo + IIV4; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.47, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

18. Primary Outcome: Mean Percentage of Perforin+CD107a- IL-2- TNF+IFNg+ CD4+ and CD8+ T Cells After Stimulation With M-001 Component Peptides
Description: as for outcome 1
Time Frame: Day 1 through Day 36
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of cells
Arm/Group | M-001 + IIV4 | Placebo + IIV4
Number analyzed (Participants) | 58 | 59
percentage of cells
  Perforin+CD107a- IL-2- TNF+IFNg+ CD4+ at Day 1 | 0.0000639 [0 to 0.000164] | 0.000372 [0.0000658 to 0.000818]
  Perforin+CD107a- IL-2- TNF+IFNg+ CD4+ Day 36 | 0 [NA to NA] — Not calculable, no cells positive for markers | 0.000485 [0.0001520 to 0.000925]
  Perforin+CD107a- IL-2- TNF+IFNg+ CD8+ Day 1 | 0.00122 [0.000315 to 0.00239] | 0.00135 [0.000376 to 0.00276]
  Perforin+CD107a- IL-2- TNF+IFNg+ CD8+ Day 36 | 0.00305 [0.001150 to 0.00542] | 0.00168 [0.000426 to 0.00360]
Statistical Analysis 1: Comparison: M-001 + IIV4 vs Placebo + IIV4; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.0061, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: M-001 + IIV4 vs Placebo + IIV4; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.28, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

19. Primary Outcome: Mean Percentage of Perforin+CD107a- IL-2- TNF+IFNg- CD4+ and CD8+ T Cells After Stimulation With M-001 Component Peptides
Description: as for outcome 1
Time Frame: Day 1 through Day 36
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of cells
Arm/Group | M-001 + IIV4 | Placebo + IIV4
Number analyzed (Participants) | 58 | 59
percentage of cells
  Perforin+CD107a- IL-2- TNF+IFNg- CD4+ at Day 1 | 0.001100 [0.000455 to 0.002030] | 0.000199 [0.0000519 to 0.000389]
  Perforin+CD107a- IL-2- TNF+IFNg- CD4+ Day 36 | 0.000564 [0.000287 to 0.000874] | 0.000454 [0.0001490 to 0.000809]
  Perforin+CD107a- IL-2- TNF+IFNg- CD8+ Day 1 | 0.00880 [0.00375 to 0.0154] | 0.00426 [0.00244 to 0.00638]
  Perforin+CD107a- IL-2- TNF+IFNg- CD8+ Day 36 | 0.00947 [0.00564 to 0.0143] | 0.00595 [0.00357 to 0.00874]
Statistical Analysis 1: Comparison: M-001 + IIV4 vs Placebo + IIV4; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.36, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: M-001 + IIV4 vs Placebo + IIV4; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.32, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

20. Primary Outcome: Mean Percentage of Perforin+CD107a- IL-2- TNF- IFNg+ CD4+ and CD8+ T Cells After Stimulation With M-001 Component Peptides
Description: as for outcome 1
Time Frame: Day 1 through Day 36
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of cells
Arm/Group | M-001 + IIV4 | Placebo + IIV4
Number analyzed (Participants) | 58 | 59
percentage of cells
  Perforin+CD107a- IL-2- TNF- IFNg+ CD4+ at Day 1 | 0.000421 [0.000135 to 0.000761] | 0.000436 [0.000198 to 0.000700]
  Perforin+CD107a- IL-2- TNF- IFNg+ CD4+ Day 36 | 0.00027 [0.0000719 to 0.000511] | 0.000438 [0.00018 to 0.000732]
  Perforin+CD107a- IL-2- TNF- IFNg+ CD8+ Day 1 | 0.00654 [0.00173 to 0.01520] | 0.00177 [0.000981 to 0.00267]
  Perforin+CD107a- IL-2- TNF- IFNg+ CD8+ Day 36 | 0.00376 [0.00151 to 0.00697] | 0.00370 [0.002230 to 0.00543]
Statistical Analysis 1: Comparison: M-001 + IIV4 vs Placebo + IIV4; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.42, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: M-001 + IIV4 vs Placebo + IIV4; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.26, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

21. Primary Outcome: Mean Percentage of Perforin+CD107a- IL-2- TNF- IFNg- CD4+ and CD8+ T Cells After Stimulation With M-001 Component Peptides
Description: as for outcome 1
Time Frame: Day 1 through Day 36
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of cells
Arm/Group | M-001 + IIV4 | Placebo + IIV4
Number analyzed (Participants) | 58 | 59
percentage of cells
  Perforin+CD107a- IL-2- TNF- IFNg- CD4+ at Day 1 | 1.180 [0.714 to 1.700] | 0.775 [0.458 to 1.140]
  Perforin+CD107a- IL-2- TNF- IFNg- CD4+ Day 36 | 1.080 [0.637 to 1.610] | 0.772 [0.475 to 1.130]
  Perforin+CD107a- IL-2- TNF- IFNg- CD8+ Day 1 | 16.0 [12.9 to 19.3] | 12.3 [10.3 to 14.4]
  Perforin+CD107a- IL-2- TNF- IFNg- CD8+ Day 36 | 16.2 [13.1 to 19.7] | 13.7 [11.3 to 16.1]
Statistical Analysis 1: Comparison: M-001 + IIV4 vs Placebo + IIV4; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.53, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: M-001 + IIV4 vs Placebo + IIV4; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.56, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

22. Primary Outcome: Mean Percentage of Perforin- CD107a+IL-2+TNF+IFNg+ CD4+ and CD8+ T Cells After Stimulation With M-001 Component Peptides
Description: as for outcome 1
Time Frame: Day 1 through Day 36
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of cells
Arm/Group | M-001 + IIV4 | Placebo + IIV4
Number analyzed (Participants) | 58 | 59
percentage of cells
  Perforin- CD107a+IL-2+TNF+IFNg+ CD4+ at Day 1 | 0.00135 [0.000809 to 0.00194] | 0.00122 [0.000714 to 0.00182]
  Perforin- CD107a+IL-2+TNF+IFNg+ CD4+ Day 36 | 0.00156 [0.000895 to 0.00229] | 0.00138 [0.00075 to 0.00211]
  Perforin- CD107a+IL-2+TNF+IFNg+ CD8+ Day 1 | 0.001170 [0.000407 to 0.00208] | 0.001000 [0.000406 to 0.001710]
  Perforin- CD107a+IL-2+TNF+IFNg+ CD8+ Day 36 | 0.000742 [0.000173 to 0.00150] | 0.000465 [0.000107 to 0.000935]
Statistical Analysis 1: Comparison: M-001 + IIV4 vs Placebo + IIV4; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.97, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: M-001 + IIV4 vs Placebo + IIV4; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.62, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

23. Primary Outcome: Mean Percentage of Perforin- CD107a+IL-2+TNF+IFNg- CD4+ and CD8+ T Cells After Stimulation With M-001 Component Peptides
Description: as for outcome 1
Time Frame: Day 1 through Day 36
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of cells
Arm/Group | M-001 + IIV4 | Placebo + IIV4
Number analyzed (Participants) | 58 | 59
percentage of cells
  Perforin- CD107a+IL-2+TNF+IFNg- CD4+ at Day 1 | 0.00230 [0.000984 to 0.00403] | 0.00200 [0.001110 to 0.00317]
  Perforin- CD107a+IL-2+TNF+IFNg- CD4+ Day 36 | 0.00212 [0.001340 to 0.00302] | 0.00144 [0.000759 to 0.00228]
  Perforin- CD107a+IL-2+TNF+IFNg- CD8+ Day 1 | 0.000197 [0 to 0.000451] | 0.0005900 [0.000134 to 0.001200]
  Perforin- CD107a+IL-2+TNF+IFNg- CD8+ Day 36 | 0.000346 [0 to 0.000801] | 0.0000719 [0 to 0.000216]
Statistical Analysis 1: Comparison: M-001 + IIV4 vs Placebo + IIV4; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.15, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: M-001 + IIV4 vs Placebo + IIV4; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.18, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

24. Primary Outcome: Mean Percentage of Perforin- CD107a+IL-2+TNF- IFNg+ CD4+ and CD8+ T Cells After Stimulation With M-001 Component Peptides
Description: as for outcome 1
Time Frame: Day 1 through Day 36
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of cells
Arm/Group | M-001 + IIV4 | Placebo + IIV4
Number analyzed (Participants) | 58 | 59
percentage of cells
  Perforin- CD107a+IL-2+TNF- IFNg+ CD4+ at Day 1 | 0 [NA to NA] — Not calculable, no cells positive for markers | 0.000156 [0 to 0.000365]
  Perforin- CD107a+IL-2+TNF- IFNg+ CD4+ Day 36 | 0.0000725 [0 to 0.000187] | 0.000078 [0 to 0.000196]
  Perforin- CD107a+IL-2+TNF- IFNg+ CD8+ Day 1 | 0 [NA to NA] — Not calculable, no cells positive for markers | 0 [NA to NA] — Not calculable, no cells positive for markers
  Perforin- CD107a+IL-2+TNF- IFNg+ CD8+ Day 36 | 0 [NA to NA] — Not calculable, no cells positive for markers | 0 [NA to NA] — Not calculable, no cells positive for markers
Statistical Analysis 1: Comparison: M-001 + IIV4 vs Placebo + IIV4; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.94, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: M-001 + IIV4 vs Placebo + IIV4; [analysis description as in outcome 1, analysis 2]; Test type: Other; No non-zero results were reported for either group so statistical testing was not performed

25. Primary Outcome: Mean Percentage of Perforin- CD107a+IL-2+TNF- IFNg- CD4+ and CD8+ T Cells After Stimulation With M-001 Component Peptides
Description: as for outcome 1
Time Frame: Day 1 through Day 36
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of cells
Arm/Group | M-001 + IIV4 | Placebo + IIV4
Number analyzed (Participants) | 58 | 59
percentage of cells
  Perforin- CD107a+IL-2+TNF- IFNg- CD4+ at Day 1 | 0.000809 [0.000198 to 0.00185] | 0.000263 [0.0000905 to 0.000468]
  Perforin- CD107a+IL-2+TNF- IFNg- CD4+ Day 36 | 0.000653 [0.000257 to 0.00114] | 0.000223 [0.0000554 to 0.000436]
  Perforin- CD107a+IL-2+TNF- IFNg- CD8+ Day 1 | 0.000377 [0.0000526 to 0.000828] | 0.000840 [0.0003060 to 0.001480]
  Perforin- CD107a+IL-2+TNF- IFNg- CD8+ Day 36 | 0.000912 [0.0002540 to 0.001770] | 0.000369 [0.0000585 to 0.000796]
Statistical Analysis 1: Comparison: M-001 + IIV4 vs Placebo + IIV4; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.14, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: M-001 + IIV4 vs Placebo + IIV4; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.26, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

26. Primary Outcome: Mean Percentage of Perforin- CD107a+IL-2- TNF+IFNg+ CD4+ and CD8+ T Cells After Stimulation With M-001 Component Peptides
Description: as for outcome 1
Time Frame: Day 1 through Day 36
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of cells
Arm/Group | M-001 + IIV4 | Placebo + IIV4
Number analyzed (Participants) | 58 | 59
percentage of cells
  Perforin- CD107a+IL-2- TNF+IFNg+ CD4+ at Day 1 | 0.00269 [0.00166 to 0.00390] | 0.00248 [0.00183 to 0.00319]
  Perforin- CD107a+IL-2- TNF+IFNg+ CD4+ Day 36 | 0.00309 [0.00206 to 0.00426] | 0.00262 [0.00171 to 0.00366]
  Perforin- CD107a+IL-2- TNF+IFNg+ CD8+ Day 1 | 0.00513 [0.00259 to 0.00834] | 0.00617 [0.00352 to 0.00921]
  Perforin- CD107a+IL-2- TNF+IFNg+ CD8+ Day 36 | 0.00604 [0.00334 to 0.00963] | 0.00374 [0.00228 to 0.00539]
Statistical Analysis 1: Comparison: M-001 + IIV4 vs Placebo + IIV4; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.72, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: M-001 + IIV4 vs Placebo + IIV4; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.31, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

27. Primary Outcome: Mean Percentage of Perforin- CD107a+IL-2- TNF+IFNg- CD4+ and CD8+ T Cells After Stimulation With M-001 Component Peptides
Description: as for outcome 1
Time Frame: Day 1 through Day 36
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of cells
Arm/Group | M-001 + IIV4 | Placebo + IIV4
Number analyzed (Participants) | 58 | 59
percentage of cells
  Perforin- CD107a+IL-2- TNF+IFNg- CD4+ at Day 1 | 0.0147 [0.00813 to 0.0239] | 0.0160 [0.01060 to 0.0230]
  Perforin- CD107a+IL-2- TNF+IFNg- CD4+ Day 36 | 0.0123 [0.00948 to 0.0153] | 0.0127 [0.00868 to 0.0177]
  Perforin- CD107a+IL-2- TNF+IFNg- CD8+ Day 1 | 0.00678 [0.00414 to 0.00986] | 0.00725 [0.00455 to 0.0104]
  Perforin- CD107a+IL-2- TNF+IFNg- CD8+ Day 36 | 0.00427 [0.00197 to 0.00726] | 0.00630 [0.00317 to 0.0107]
Statistical Analysis 1: Comparison: M-001 + IIV4 vs Placebo + IIV4; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.31, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: M-001 + IIV4 vs Placebo + IIV4; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.22, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

28. Primary Outcome: Mean Percentage of Perforin- CD107a+IL-2- TNF- IFNg+ CD4+ and CD8+ T Cells After Stimulation With M-001 Component Peptides
Description: as for outcome 1
Time Frame: Day 1 through Day 36
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of cells
Arm/Group | M-001 + IIV4 | Placebo + IIV4
Number analyzed (Participants) | 58 | 59
percentage of cells
  Perforin- CD107a+IL-2- TNF- IFNg+ CD4+ at Day 1 | 0.000511 [0.000253 to 0.000815] | 0.000694 [0.000345 to 0.001090]
  Perforin- CD107a+IL-2- TNF- IFNg+ CD4+ Day 36 | 0.000731 [0.000391 to 0.001110] | 0.001910 [0.000921 to 0.003160]
  Perforin- CD107a+IL-2- TNF- IFNg+ CD8+ Day 1 | 0.001580 [0.000815 to 0.002530] | 0.002160 [0.001100 to 0.003380]
  Perforin- CD107a+IL-2- TNF- IFNg+ CD8+ Day 36 | 0.001780 [0.000916 to 0.002790] | 0.002240 [0.001290 to 0.003310]
Statistical Analysis 1: Comparison: M-001 + IIV4 vs Placebo + IIV4; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.16, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: M-001 + IIV4 vs Placebo + IIV4; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.44, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

29. Primary Outcome: Mean Percentage of Perforin- CD107a+IL-2- TNF- IFNg- CD4+ and CD8+ T Cells After Stimulation With M-001 Component Peptides
Description: as for outcome 1
Time Frame: Day 1 through Day 36
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of cells
Arm/Group | M-001 + IIV4 | Placebo + IIV4
Number analyzed (Participants) | 58 | 59
percentage of cells
  Perforin- CD107a+IL-2- TNF- IFNg- CD4+ at Day 1 | 0.231 [0.178 to 0.292] | 0.240 [0.179 to 0.314]
  Perforin- CD107a+IL-2- TNF- IFNg- CD4+ Day 36 | 0.220 [0.172 to 0.277] | 0.236 [0.184 to 0.293]
  Perforin- CD107a+IL-2- TNF- IFNg- CD8+ Day 1 | 0.294 [0.226 to 0.374] | 0.323 [0.237 to 0.434]
  Perforin- CD107a+IL-2- TNF- IFNg- CD8+ Day 36 | 0.295 [0.232 to 0.366] | 0.341 [0.267 to 0.424]
Statistical Analysis 1: Comparison: M-001 + IIV4 vs Placebo + IIV4; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.67, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: M-001 + IIV4 vs Placebo + IIV4; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.48, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

30. Primary Outcome: Mean Percentage of Perforin- CD107a- IL-2+TNF+IFNg+ CD4+ and CD8+ T Cells After Stimulation With M-001 Component Peptides
Description: as for outcome 1
Time Frame: Day 1 through Day 36
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of cells
Arm/Group | M-001 + IIV4 | Placebo + IIV4
Number analyzed (Participants) | 58 | 59
percentage of cells
  Perforin- CD107a- IL-2+TNF+IFNg+ CD4+ at Day 1 | 0.00328 [0.00238 to 0.00430] | 0.00365 [0.00230 to 0.00548]
  Perforin- CD107a- IL-2+TNF+IFNg+ CD4+ Day 36 | 0.00955 [0.00604 to 0.01470] | 0.00289 [0.00201 to 0.00390]
  Perforin- CD107a- IL-2+TNF+IFNg+ CD8+ Day 1 | 0.000238 [0 to 0.000657] | 0.000693 [0.0000839 to 0.001620]
  Perforin- CD107a- IL-2+TNF+IFNg+ IFNg- CD8+ Day 36 | 0.000288 [0.0000404 to 0.000626] | 0.000486 [0 to 0.001300]
Statistical Analysis 1: Comparison: M-001 + IIV4 vs Placebo + IIV4; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: M-001 + IIV4 vs Placebo + IIV4; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.62, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

31. Primary Outcome: Mean Percentage of Perforin- CD107a- IL-2+TNF+IFNg- CD4+ and CD8+ T Cells After Stimulation With M-001 Component Peptides
Description: as for outcome 1
Time Frame: Day 1 through Day 36
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of cells
Arm/Group | M-001 + IIV4 | Placebo + IIV4
Number analyzed (Participants) | 58 | 59
percentage of cells
  Perforin- CD107a- IL-2+TNF+IFNg- CD4+ at Day 1 | 0.01170 [0.00784 to 0.01600] | 0.01240 [0.00958 to 0.01540]
  Perforin- CD107a- IL-2+TNF+IFNg- CD4+ Day 36 | 0.01640 [0.01230 to 0.02130] | 0.01130 [0.00789 to 0.01540]
  Perforin- CD107a- IL-2+TNF+IFNg- CD8+ Day 1 | 0.00161 [0.000488 to 0.00318] | 0.00184 [0.000851 to 0.00301]
  Perforin- CD107a- IL-2+TNF+IFNg- IFNg- CD8+ Day 36 | 0.00129 [0.000535 to 0.00224] | 0.00102 [0.000354 to 0.00186]
Statistical Analysis 1: Comparison: M-001 + IIV4 vs Placebo + IIV4; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.0093, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: M-001 + IIV4 vs Placebo + IIV4; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.51, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

32. Primary Outcome: Mean Percentage of Perforin- CD107a- IL-2+TNF- IFNg+ CD4+ and CD8+ T Cells After Stimulation With M-001 Component Peptides
Description: as for outcome 1
Time Frame: Day 1 through Day 36
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of cells
Arm/Group | M-001 + IIV4 | Placebo + IIV4
Number analyzed (Participants) | 58 | 59
percentage of cells
  Perforin- CD107a- IL-2+TNF- IFNg+ CD4+ at Day 1 | 0.000169 [0.0000294 to 0.000355] | 0.000438 [0.000195 to 0.000714]
  Perforin- CD107a- IL-2+TNF- IFNg+ CD4+ Day 36 | 0.000434 [0.0001960 to 0.000702] | 0.000372 [0.000131 to 0.000680]
  Perforin- CD107a- IL-2+TNF- IFNg+ CD8+ Day 1 | 0.000397 [0 to 0.000977] | 0.000339 [0.0000652 to 0.000709]
  Perforin- CD107a- IL-2+TNF- IFNg+ CD8+ Day 36 | 0.000487 [0 to 0.001360] | 0.000378 [0.0000775 to 0.000736]
Statistical Analysis 1: Comparison: M-001 + IIV4 vs Placebo + IIV4; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.54, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: M-001 + IIV4 vs Placebo + IIV4; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.43, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

33. Primary Outcome: Mean Percentage of Perforin- CD107a- IL-2+TNF- IFNg- CD4+ and CD8+ T Cells After Stimulation With M-001 Component Peptides
Description: as for outcome 1
Time Frame: Day 1 through Day 36
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of cells
Arm/Group | M-001 + IIV4 | Placebo + IIV4
Number analyzed (Participants) | 58 | 59
percentage of cells
  Perforin- CD107a- IL-2+TNF- IFNg- CD4+ at Day 1 | 0.0445 [0.0285 to 0.0625] | 0.0400 [0.0283 to 0.0530]
  Perforin- CD107a- IL-2+TNF- IFNg- CD4+ Day 36 | 0.0395 [0.0274 to 0.0524] | 0.0478 [0.0343 to 0.0627]
  Perforin- CD107a- IL-2+TNF- IFNg- CD8+ Day 1 | 0.0468 [0.0311 to 0.0645] | 0.0444 [0.0310 to 0.0605]
  Perforin- CD107a- IL-2+TNF- IFNg- CD8+ Day 36 | 0.0417 [0.0272 to 0.0588] | 0.0522 [0.0402 to 0.0653]
Statistical Analysis 1: Comparison: M-001 + IIV4 vs Placebo + IIV4; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.44, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: M-001 + IIV4 vs Placebo + IIV4; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.014, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

34. Primary Outcome: Mean Percentage of Perforin- CD107a- IL-2- TNF+IFNg+ CD4+ and CD8+ T Cells After Stimulation With M-001 Component Peptides
Description: as for outcome 1
Time Frame: Day 1 through Day 36
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of cells
Arm/Group | M-001 + IIV4 | Placebo + IIV4
Number analyzed (Participants) | 58 | 59
percentage of cells
  Perforin- CD107a- IL-2- TNF+IFNg+ CD4+ at Day 1 | 0.00935 [0.00716 to 0.01180] | 0.00881 [0.00622 to 0.01190]
  Perforin- CD107a- IL-2- TNF+IFNg+ CD4+ Day 36 | 0.01520 [0.01160 to 0.01950] | 0.00731 [0.00556 to 0.00926]
  Perforin- CD107a- IL-2- TNF+IFNg+ CD8+ Day 1 | 0.00488 [0.00305 to 0.00702] | 0.00460 [0.00242 to 0.00751]
  Perforin- CD107a- IL-2- TNF+IFNg+CD8+ Day 36 | 0.00257 [0.00141 to 0.00398] | 0.00242 [0.00139 to 0.00357]
Statistical Analysis 1: Comparison: M-001 + IIV4 vs Placebo + IIV4; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: M-001 + IIV4 vs Placebo + IIV4; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.96, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

35. Primary Outcome: Mean Percentage of Perforin- CD107a- IL-2- TNF+IFNg- CD4+ and CD8+ T Cells After Stimulation With M-001 Component Peptides
Description: as for outcome 1
Time Frame: Day 1 through Day 36
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of cells
Arm/Group | M-001 + IIV4 | Placebo + IIV4
Number analyzed (Participants) | 58 | 59
percentage of cells
  Perforin- CD107a- IL-2- TNF+IFNg- CD4+ at Day 1 | 0.390 [0.288 to 0.508] | 0.483 [0.331 to 0.669]
  Perforin- CD107a- IL-2- TNF+IFNg- CD4+ Day 36 | 0.389 [0.280 to 0.524] | 0.354 [0.263 to 0.459]
  Perforin- CD107a- IL-2- TNF+IFNg- CD8+ Day 1 | 0.0388 [0.0201 to 0.0676] | 0.0415 [0.0254 to 0.0618]
  Perforin- CD107a- IL-2- TNF+IFNg- CD8+ Day 36 | 0.0341 [0.0175 to 0.0613] | 0.0348 [0.0227 to 0.0503]
Statistical Analysis 1: Comparison: M-001 + IIV4 vs Placebo + IIV4; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.65, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: M-001 + IIV4 vs Placebo + IIV4; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.53, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

36. Primary Outcome: Mean Percentage of Perforin- CD107a- IL-2- TNF- IFNg+ CD4+ and CD8+ T Cells After Stimulation With M-001 Component Peptides
Description: as for outcome 1
Time Frame: Day 1 through Day 36
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of cells
Arm/Group | M-001 + IIV4 | Placebo + IIV4
Number analyzed (Participants) | 58 | 59
percentage of cells
  Perforin- CD107a- IL-2- TNF- IFNg+ CD4+ at Day 1 | 0.0238 [0.0164 to 0.0354] | 0.0147 [0.0119 to 0.0178]
  Perforin- CD107a- IL-2- TNF- IFNg+ CD4+ Day 36 | 0.0199 [0.0155 to 0.0252] | 0.0255 [0.0133 to 0.0466]
  Perforin- CD107a- IL-2- TNF- IFNg+ CD8+ Day 1 | 0.0314 [0.0165 to 0.0505] | 0.0209 [0.0131 to 0.0307]
  Perforin- CD107a- IL-2- TNF- IFNg+ CD8+ Day 36 | 0.0318 [0.0200 to 0.0467] | 0.0308 [0.0180 to 0.0473]
Statistical Analysis 1: Comparison: M-001 + IIV4 vs Placebo + IIV4; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.35, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: M-001 + IIV4 vs Placebo + IIV4; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.66, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

37. Primary Outcome: Mean Percentage of Perforin- CD107a- IL-2- TNF- IFNg- CD4+ and CD8+ T Cells After Stimulation With M-001 Component Peptides
Description: as for outcome 1
Time Frame: Day 1 through Day 36
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of cells
Arm/Group | M-001 + IIV4 | Placebo + IIV4
Number analyzed (Participants) | 58 | 59
percentage of cells
  Perforin- CD107a- IL-2- TNF- IFNg- CD4+ at Day 1 | 98.1 [97.5 to 98.6] | 98.4 [98.0 to 98.8]
  Perforin- CD107a- IL-2- TNF- IFNg- CD4+ Day 36 | 98.2 [97.6 to 98.7] | 98.5 [98.2 to 98.8]
  Perforin- CD107a- IL-2- TNF- IFNg- CD8+ Day 1 | 83.5 [80.2 to 86.6] | 87.2 [85.1 to 89.1]
  Perforin- CD107a- IL-2- TNF- IFNg- CD8+ Day 36 | 83.2 [79.8 to 86.5] | 85.8 [83.3 to 88.2]
Statistical Analysis 1: Comparison: M-001 + IIV4 vs Placebo + IIV4; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.86, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: M-001 + IIV4 vs Placebo + IIV4; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.53, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

38. Primary Outcome: Number of Participants With Clinical Safety Laboratory Adverse Events After the First M-001 Vaccination
Description: Blood was collected after first vaccination for assessment by a central clinical laboratory. Clinical safety laboratory adverse events included white blood cells (WBC) </=3900/uL or >/=10,600/uL; platelets </=139,000/uL or >/=416,000/uL; hemoglobin </=11.4 g/dL (female) or </=12.4 g/dL (male); alanine aminotransferase (ALT) >/=44 IU/L (female) or >/=61 IU/L (male); creatinine >/=1.1 mg/dL (female) or >/=1.4 (male); and total bilirubin >/=1.30 mg/dL.
Time Frame: Day 9
Population: The Safety Analysis population includes all participants who received the first dose of study product and have a result reported for the parameter.
Measure: Count of Participants; unit: Participants
Arm/Group | M-001 + IIV4 | Placebo + IIV4
Number analyzed (Participants) | 61 | 59
Participants
  WBC | 5 | 7
  platelets: number analyzed (Participants) | 60 | 59
  platelets | 1 | 0
  hemoglobin | 3 | 1
  ALT | 2 | 0
  creatinine | 0 | 0
  total bilirubin: number analyzed (Participants) | 60 | 58
  total bilirubin | 2 | 2

39. Primary Outcome: Number of Participants With Clinical Safety Laboratory Adverse Events After Second M-001 Vaccination
Description: Clinical safety laboratory adverse events included WBC less than or equal to 3900/uL or greater than or equal to 10,600/uL; platelets less than or equal to 139,000/uL or greater than or equal to 416,000/uL; hemoglobin less than or equal to 11.4 g/dL (female) or less than or equal to 12.4 g/dL (male); alanine aminotransferase (ALT) greater than or equal to 44 IU/L (female) or greater than or equal to 61 IU/L (male); creatinine greater than or equal to 1.1 mg/dL (female) or greater than or equal to 1.4 (male); and total bilirubin greater than or equal to 1.30 mg/dL.
Time Frame: Day 22 through Day 29
Population: The Safety Analysis population includes all participants who received the second dose of study product and have a result reported for the parameter.
Measure: Count of Participants; unit: Participants
Arm/Group | M-001 + IIV4 | Placebo + IIV4
Number analyzed (Participants) | 54 | 55
Participants
  WBC | 2 | 3
  platelets: number analyzed (Participants) | 53 | 55
  platelets | 0 | 0
  hemoglobin | 2 | 0
  ALT | 2 | 0
  creatinine | 0 | 0
  total bilirubin: number analyzed (Participants) | 52 | 54
  total bilirubin | 2 | 2

40. Primary Outcome: Number of Participants Reporting Solicited Injection Site and Systemic Reactogenicity Events After the First M-001 Vaccination
Description: Participants maintained a memory aid and thermometer to record daily oral temperatures and the occurrence of systemic reactions of feverishness, fatigue, malaise, myalgia, arthralgia, headache, and nausea, as well as local injection site reactions of pain, tenderness, redness, and swelling for 8 days after vaccination (Day 0-7) based on their interference with daily activities, with a severity grade of mild meaning no interference, moderate as some interference and severe as significant interference/prevented daily activity. Fever was defined as an oral temperature of 38 degree Celsius or higher. Participants are counted if they reported experiencing the symptom at any severity on any of the 8 days post vaccination.
Time Frame: Day 1 through Day 8
Population: The Safety Analysis population includes all participants who received the first study product.
Measure: Count of Participants; unit: Participants
Arm/Group | M-001 + IIV4 | Placebo + IIV4
Number analyzed (Participants) | 61 | 59
Participants
  Fever | 0 | 1
  Feverishness | 1 | 3
  Fatigue | 14 | 14
  Malaise | 5 | 5
  Myalgia | 6 | 6
  Arthralgia | 1 | 1
  Headache | 13 | 15
  Nausea | 7 | 1
  Injection site pain | 12 | 2
  Injection site tenderness | 24 | 9
  Injection site itchiness/pruritus | 2 | 1
  Injection site ecchymosis | 2 | 3
  Injection site erythema | 14 | 11
  Injection site induration/swelling | 3 | 4

41. Primary Outcome: Number of Participants Reporting Solicited Injection Site and Systemic Reactogenicity Events After the Second M-001 Vaccination
Description: as for outcome 40
Time Frame: Day 22 through Day 29
Population: The Safety Analysis population includes all participants who received the second study product.
Measure: Count of Participants; unit: Participants
Arm/Group | M-001 + IIV4 | Placebo + IIV4
Number analyzed (Participants) | 55 | 55
Participants
  Fever | 1 | 0
  Feverishness | 1 | 2
  Fatigue | 8 | 7
  Malaise | 6 | 4
  Myalgia | 4 | 2
  Arthralgia | 0 | 2
  Headache | 8 | 8
  Nausea | 2 | 1
  Injection site pain | 13 | 2
  Injection site tenderness | 16 | 11
  Injection site itchiness/pruritus | 2 | 1
  Injection site ecchymosis | 0 | 3
  Injection site erythema | 15 | 7
  Injection site induration/swelling | 2 | 2

42. Primary Outcome: Number of Participants Reporting Vaccine-related Serious Adverse Events (SAEs) After M-001 Vaccination
Description: SAEs included any untoward medical occurrence that resulted in death; was life threatening; was a persistent/significant disability/incapacity; required inpatient hospitalization or prolongation or a congenital anomaly/birth defect. Relationship (related or unrelated to the study product) was determined by a site principal investigator blinded to the study product received by the participant.
Time Frame: Day 1 through Day 200
Population: The Safety Analysis population includes all participants who received at least one dose of study product.
Measure: Count of Participants; unit: Participants
Arm/Group | M-001 + IIV4 | Placebo + IIV4
Number analyzed (Participants) | 61 | 59
Participants | 0 | 0

43. Secondary Outcome: Number of Participants Reporting Serious Adverse Events (SAEs) After M-001 Vaccination
Description: SAEs included any untoward medical occurrence that resulted in death; was life threatening; was a persistent/significant disability/incapacity; required inpatient hospitalization or prolongation or a congenital anomaly/birth defect. All events are included regardless of relationship to the study product.
Time Frame: Day 1 through Day 200
Population: The Safety Analysis population includes all participants who received at least one dose of study product.
Measure: Count of Participants; unit: Participants
Arm/Group | M-001 + IIV4 | Placebo + IIV4
Number analyzed (Participants) | 61 | 59
Participants | 1 | 0

44. Secondary Outcome: Incidence of Unsolicited Non-serious Adverse Events (AEs) After M-001 Vaccination
Description: Unsolicited adverse events were collected from the time of first vaccination and at each follow-up visit through Day 43. Adverse events were defined as any untoward medical occurrence regardless of its causal relationship to the study treatment. Events were coded with MedDRA and are reported by System Organ Class.
Time Frame: Day 1 through Day 43
Population: The Safety Analysis population includes all participants who received at least one dose of study product.
Measure: Number; unit: participants
Arm/Group | M-001 + IIV4 | Placebo + IIV4
Number analyzed (Participants) | 61 | 59
participants
  Blood and lymphatic system disorders | 0 | 2
  Eye Disorders | 1 | 1
  Gastrointestinal disorders | 2 | 1
  Immune system disorders | 0 | 1
  Infections and Infestations | 11 | 12
  Injury, poisoning and procedural complications | 2 | 2
  Musculoskeletal and connective tissue disorders | 4 | 1
  Nervous system disorders | 3 | 2
  Reproductive system and breast disorders | 1 | 0
  Respiratory, thoracic and mediastinal disorders | 3 | 2
  Skin and subcutaneous tissue disorders | 3 | 3
  Vascular disorders | 0 | 1

45. Secondary Outcome: The Percentage of Subjects Achieving HAI Seroconversion to IIV4 Vaccine Virus From Day 172 to Day 200
Description: Blood was collected from participants for testing in the HAI assay with the vaccine viruses as the assay antigens. Seroconversion was defined as a Day 172 titer less than 10 and Day 200 titer greater than or equal to 40, or for those with a Day 172 titer of 10 or greater, a minimum 4-fold rise in Day 200 antibody titer.
Time Frame: Day 172 to Day 200
Population: The modified intent-to-treat (mITT) population includes all participants who received at least one dose of study vaccine and contributed at least one post-study vaccination venous blood sample for immunogenicity testing for which valid results were reported
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | M-001 + IIV4 | Placebo + IIV4
Number analyzed (Participants) | 52 | 50
percentage of participants
  B/Colorado/6/2017 | 13.5 [5.6 to 25.8] | 6.0 [1.3 to 16.5]
  B/Phuket/3073/2013 | 11.5 [4.4 to 23.4] | 8.0 [2.2 to 19.2]
  A/Michigan/45/2015 X-275 | 15.4 [6.9 to 28.1] | 16.0 [7.2 to 29.1]
  A/Singapore/INFIMH-16-0019/2016 NIB-104 | 25.0 [14.0 to 38.9] | 20.0 [10.0 to 33.7]

46. Secondary Outcome: The Percentage of Subjects Achieving Neutralizing Antibody Seroconversion to IIV4 Vaccine Virus From Day 172 to Day 200
Description: Blood was collected from participants for testing in the neutralizing antibody assay with the vaccine viruses as the assay antigens. Seroconversion was defined as a Day 172 titer less than 10 and Day 200 titer greater than or equal to 40, or for those with a Day 172 titer of 10 or greater, a minimum 4-fold rise in Day 200 antibody titer.
Time Frame: Day 172 to Day 200
Population: as for outcome 45
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | M-001 + IIV4 | Placebo + IIV4
Number analyzed (Participants) | 52 | 50
percentage of participants
  B/Colorado/6/2017 | 17.3 [8.2 to 30.3] | 6.0 [1.3 to 16.5]
  B/Phuket/3073/2013 | 13.5 [5.6 to 25.8] | 8.0 [2.2 to 19.2]
  A/Michigan/45/2015 X-275 | 19.2 [9.6 to 32.5] | 16.0 [7.2 to 29.1]
  A/Singapore/INFIMH-16-0019/2016 NIB-104 | 46.2 [32.2 to 60.5] | 26.0 [14.6 to 40.3]

47. Secondary Outcome: The Percentage of Participants With an HAI Antibody Titer of 40 or Greater and GMTs vs. IIV4 Vaccine Viruses at Day 1
Description: Blood was collected from participants for testing in the HAI assay with the vaccine viruses as the assay antigens. Each sample was tested at least twice according to standard operating procedures and the result of each replicate reported. A participant is counted if the geometric mean of the replicate values was 40 or greater.
Time Frame: Day 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | M-001 + IIV4 | Placebo + IIV4
Number analyzed (Participants) | 55 | 55
percentage of participants
  B/Colorado/6/2017 | 98.3 [91.1 to 100] | 93.2 [83.5 to 98.1]
  B/Phuket/3073/2013 | 93.3 [83.8 to 98.2] | 93.2 [83.5 to 98.1]
  A/Michigan/45/2015 X-275 | 80.0 [67.7 to 89.2] | 81.4 [69.1 to 90.3]
  A/Singapore/INFIMH-16-0019/2016 NIB-104 | 43.3 [30.6 to 56.8] | 33.9 [22.1 to 47.4]

48. Secondary Outcome: The Percentage of Participants With an HAI Antibody Titer of 40 or Greater and GMTs vs. IIV4 Vaccine Viruses at Day 43
Description: as for outcome 47
Time Frame: Day 43
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | M-001 + IIV4 | Placebo + IIV4
Number analyzed (Participants) | 53 | 53
percentage of participants
  B/Colorado/6/2017 | 96.2 [87.0 to 99.5] | 92.5 [81.8 to 97.9]
  B/Phuket/3073/2013 | 94.3 [84.3 to 98.8] | 92.5 [81.8 to 97.9]
  A/Michigan/45/2015 X-275 | 79.2 [65.9 to 89.2] | 79.2 [65.9 to 89.2]
  A/Singapore/INFIMH-16-0019/2016 NIB-104 | 39.6 [26.5 to 54.0] | 35.8 [23.1 to 50.2]

49. Secondary Outcome: The Percentage of Participants With an HAI Antibody Titer of 40 or Greater and GMTs vs. IIV4 Vaccine Viruses at Day 172
Description: as for outcome 47
Time Frame: Day 172
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | M-001 + IIV4 | Placebo + IIV4
Number analyzed (Participants) | 53 | 52
percentage of participants
  B/Colorado/6/2017 | 94.3 [84.3 to 98.8] | 88.5 [76.6 to 95.6]
  B/Phuket/3073/2013 | 94.3 [84.3 to 98.8] | 88.5 [76.6 to 95.6]
  A/Michigan/45/2015 X-275 | 81.1 [68.0 to 90.6] | 78.8 [65.3 to 88.9]
  A/Singapore/INFIMH-16-0019/2016 NIB-104 | 39.6 [26.5 to 54.0] | 30.8 [18.7 to 45.1]

50. Secondary Outcome: The Percentage of Participants With an HAI Antibody Titer of 40 or Greater and GMTs vs. IIV4 Vaccine Viruses at Day 200
Description: as for outcome 47
Time Frame: Day 200
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | M-001 + IIV4 | Placebo + IIV4
Number analyzed (Participants) | 52 | 50
percentage of participants
  B/Colorado/6/2017 | 98.1 [89.7 to 100] | 96.0 [86.3 to 99.5]
  B/Phuket/3073/2013 | 98.1 [89.7 to 100] | 96.0 [86.3 to 99.5]
  A/Michigan/45/2015 X-275 | 94.2 [84.1 to 98.8] | 88.0 [75.7 to 95.5]
  A/Singapore/INFIMH-16-0019/2016 NIB-104 | 67.3 [52.9 to 79.7] | 60 [45.2 to 73.6]

51. Secondary Outcome: The Percentage of Participants With a Neutralizing Antibody Titer of 40 or Greater and GMTs vs. IIV4 Vaccine Viruses at Day 1
Description: Blood was collected from participants for testing in the neutralizing antibody assay with the vaccine viruses as the assay antigens. Each sample was tested at least twice according to standard operating procedures and the result of each replicate reported. A participant is counted if the geometric mean of the replicate values was 40 or greater.
Time Frame: Day 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | M-001 + IIV4 | Placebo + IIV4
Number analyzed (Participants) | 60 | 59
percentage of participants
  B/Colorado/6/2017 | 30.0 [18.8 to 43.2] | 22.0 [12.3 to 34.7]
  B/Phuket/3073/2013 | 71.7 [58.6 to 82.5] | 74.6 [61.6 to 85.0]
  A/Michigan/45/2015 X-275 | 100 [94.0 to 100] | 96.6 [88.3 to 99.6]
  A/Singapore/INFIMH-16-0019/2016 NIB-104 | 91.7 [81.6 to 97.2] | 93.2 [83.5 to 989.1]

52. Secondary Outcome: The Percentage of Participants With a Neutralizing Antibody Titer of 40 or Greater and GMTs vs. IIV4 Vaccine Viruses at Day 43
Description: as for outcome 51
Time Frame: Day 43
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | M-001 + IIV4 | Placebo + IIV4
Number analyzed (Participants) | 53 | 53
percentage of participants
  B/Colorado/6/2017 | 20.8 [10.8 to 34.1] | 28.3 [16.8 to 42.3]
  B/Phuket/3073/2013 | 77.4 [63.8 to 87.7] | 69.8 [55.7 to 81.7]
  A/Michigan/45/2015 X-275 | 98.1 [89.9 to 100] | 98.1 [89.9 to 100]
  A/Singapore/INFIMH-16-0019/2016 NIB-104 | 90.6 [79.3 to 96.9] | 92.5 [81.8 to 97.9]

53. Secondary Outcome: The Percentage of Participants With a Neutralizing Antibody Titer of 40 or Greater and GMTs vs. IIV4 Vaccine Viruses at Day 172
Description: as for outcome 51
Time Frame: Day 172
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | M-001 + IIV4 | Placebo + IIV4
Number analyzed (Participants) | 53 | 52
percentage of participants
  B/Colorado/6/2017 | 24.5 [13.8 to 38.3] | 26.9 [15.6 to 41.0]
  B/Phuket/3073/2013 | 67.9 [53.7 to 80.1] | 69.2 [54.9 to 81.3]
  A/Michigan/45/2015 X-275 | 98.1 [89.9 to 100] | 96.2 [86.8 to 99.5]
  A/Singapore/INFIMH-16-0019/2016 NIB-104 | 86.8 [74.7 to 94.5] | 92.3 [81.5 to 97.9]

54. Secondary Outcome: The Percentage of Participants With a Neutralizing Antibody Titer of 40 or Greater and GMTs vs. IIV4 Vaccine Viruses at Day 200
Description: as for outcome 51
Time Frame: Day 200
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | M-001 + IIV4 | Placebo + IIV4
Number analyzed (Participants) | 52 | 50
percentage of participants
  B/Colorado/6/2017 | 69.2 [54.9 to 81.3] | 50.0 [35.5 to 64.5]
  B/Phuket/3073/2013 | 86.5 [74.2 to 94.4] | 82.0 [68.6 to 91.4]
  A/Michigan/45/2015 X-275 | 100 [93.2 to 100] | 100 [92.9 to 100]
  A/Singapore/INFIMH-16-0019/2016 NIB-104 | 98.1 [89.7 to 100] | 98.0 [89.4 to 99.9]

ADVERSE EVENTS:
Time Frame: Solicited events were collected for 8 days after each vaccination, unsolicited non-serious AEs through 28 days after the second study vaccination, and SAEs through approximately Day 200.
Description: For events solicited on the Memory Aid in the 8 days after vaccination, a participant was considered to have one event if it was reported as experienced at any time in the 8-day period. Each 8-day period was considered a separate event.
Arm/Group | M-001 + IIV4 | Placebo + IIV4
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/59
Serious Adverse Events (participants affected / at risk) | 1/61 | 0/59
Other Adverse Events (participants affected / at risk) | 52/61 | 44/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | M-001 + IIV4 (N=61) | Placebo + IIV4 (N=59)
Deafness (Ear and labyrinth disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | M-001 + IIV4 (N=61) | Placebo + IIV4 (N=59)
Respiratory Tract Infection (Infections and infestations) | 3 (3) | 5 (5)
Nausea (Gastrointestinal disorders) | 9 (9) | 1 (2)
Fatigue (General disorders) | 18 (22) | 16 (21)
Feeling Hot (General disorders) | 2 (2) | 4 (5) — Solicited as 'feverishness'
Injection Site Erythema (General disorders) | 22 (29) | 14 (18)
Injection Site Haemorrhage (General disorders) | 2 (2) | 5 (6)
Injection Site Induration (General disorders) | 5 (5) | 5 (6)
Injection Site Pain (General disorders) | 33 (46) | 14 (20)
Malaise (General disorders) | 9 (11) | 7 (9)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 9 (10) | 7 (8)
Headache (Nervous system disorders) | 17 (21) | 18 (23)
Blood Bilirubin Increased (Investigations) | 2 (4) | 3 (4)
Haemoglobin Decreased (Investigations) | 5 (6) | 1 (1)
White Blood Cell Count Decreased (Investigations) | 3 (4) | 5 (5)
White Blood Cell Count Increased (Investigations) | 4 (4) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-09-09): https://cdn.clinicaltrials.gov/large-docs/92/NCT03058692/SAP_000.pdf
  • Study Protocol (2018-12-06): https://cdn.clinicaltrials.gov/large-docs/92/NCT03058692/Prot_001.pdf